CLINICAL TRIAL: NCT05027113
Title: App-Based Mindfulness Meditation for People of Color Who Experience Race-Related Stress: A Randomized Control Trial
Brief Title: App-Based Mindfulness Meditation for People of Color Who Experience Race-Related Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Giovanni Ramos, MA, CPhil, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-005750
Record Dates: First submitted 2021-08-13; First posted 2021-08-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stress, Psychological; Anxiety; Depression; Rumination; Emotional Regulation; Mindfulness; Self-Compassion; Emotional Distress
Keywords: Race-Related Stress; Mental Health; Mindfulness; Meditation; App
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; Rumination Syndrome; Emotional Regulation; Psychological Well-Being; Alzheimer Disease | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Individuals who meet eligibility criteria will be randomized to either the intervention group (n = 40) or a wait-list control group (n = 40),
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be aware of whether they were randomized to the intervention group or the wait-list control group. The intervention is self-guided and automated through the use of a smartphone app. As such, masking is not an issue. The principal investigator will not be involved with randomization. Assessments are self-administered via online questionnaires. As such, masking is not relevant in terms of outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Us (Experimental): Use of the 10% Happier app to complete at least one meditation daily -with the possibility of exceeding this goal by choosing additional meditations- for 4 weeks. Participants will be asked to complete "The Basics" and "The Basics II" courses to familiarize themselves with the principles of mindfulness meditation. Each audio-recorded session begins with a short video providing psychoeducation around mindfulness meditation and teaching specific techniques (e.g., using the breath as an anchor, redirecting attention, noting thoughts and emotions). For the last two weeks of the program, participants will be invited to complete the "Essential Advice" course. This additional course is composed of 14 sessions ranging in length from 15 to 18 minutes.
  Interventions: Behavioral: Mindfulness meditation
- Assessments First (No Intervention): Wait-list control group. Individuals in this group will complete baseline, mid-, and post-treatment assessments before receiving the intervention (i.e., 4 weeks after randomization).

INTERVENTIONS:
Behavioral: Mindfulness meditation — Participants use the meditation app 10% Happier to practice mindfulness meditation (see detailed description in arm/group section)
  Other Names: Mind-Us
  Arms: Mind-Us

SUMMARY:
In the United States, people of color (POC) are disproportionally affected by stressors related to race/ethnicity compared with their non-Latinx White (NLW). Considering POC exposed to race-related stress are at high risk of developing a mental health disorder, there is a clear need for treatments that allow individuals to cope effectively with these stressors.

Among many evidence-based treatments available, mindfulness-based interventions (MBIs) may be particularly well suited to help POC cope. MBIs are hypothesized to be effective via increases in mindfulness and self-compassion, as well as reductions in experiential avoidance, rumination, and emotion suppression. Despite their effectiveness, MBIs rarely reach POC. As such, innovative strategies such as self-directed app-based intervention may reduce the treatment gap.

Considering the lack of research examining the effectiveness of MBIs among POC, especially those who experience elevated levels of race-related stress, this study will employ a randomized control trial (RCT) approach to examine whether receiving an app-based MBI engages the hypothesized mechanisms of change (i.e., mindfulness, self-compassion, experiential avoidance, rumination, emotion suppression) among POC. Similarly, the study will test whether the intervention leads to decreases in the negative mental health outcomes more often associated with exposure to race-related stress (i.e., stress, anxiety, depression). Acceptability, adherence, and satisfaction also will be analyzed to explore whether a non-culturally adapted MBI is still relevant for POC who face race-related stress. Results from this trial will contribute to the nascent data on MBI acceptability and effectiveness with POC. To the investigators' knowledge, this study will also be the first to include a sample of POC recruited based on elevated levels of race-related stress, a high-risk population that is not commonly targeted in MBI research.

DETAILED DESCRIPTION:
In the United States, people of color (POC) are disproportionally affected by stressors related to race/ethnicity compared with their non-Latinx White (NLW) counterparts, with approximately 70% of POC reporting having experienced some form of discrimination in their lives and 60% reporting facing day-to-day discriminatory treatment. Race-related stress is the psychological distress associated with appraising a situation as disturbing or burdensome because of negative racial bias. Race-related stressors have multiple forms, such as direct interpersonal discrimination (i.e., perceived differential and unfair treatment among individuals), vicarious discrimination (i.e., observing members of one's race/ethnicity being victimized), institutional practices (i.e., laws and policies that limit access to services and opportunities), and cultural traditions (i.e., beliefs and practices that reinforce the idea of NLW's superiority over POC).

When differential or unfair treatment is perceived, it triggers physiological (e.g., cardiovascular reactivity, dysregulated HPA axis activity), cognitive-affective (e.g., rumination, emotion suppression), and behavioral (e.g., avoidance, aggression) responses that prepare the individual to confront the situation. Although this acute stress response may be beneficial in the short term, the chronic and unpredictable nature of race-related stressors often depletes an individual's psychological resources and increases their vulnerability to developing mental health disorders. Metanalytic work supports this stress-response model among POC, showing that exposure to race-related stress is a consistent predictor of increases in mental health problems, including overall stress, anxiety, and depressive symptoms.

Among many EBTs available, mindfulness-based interventions (MBIs) may be particularly well suited to achieve these goals. Mindfulness is a psychological trait associated with staying in the present moment with one's experience (i.e., physical sensations, thoughts, emotions, behaviors), endorsing a nonjudgmental and curious attitude, and cultivating acceptance and self-compassion. Self-compassion refers to an attitude of openness to one's own suffering without avoiding it, cultivating the desire to alleviate it without self-judgment. In MBIs, participants cultivate these two qualities through meditations -exercises aimed to gain awareness of one's experience with an accepting and compassionate attitude. Metanalyses show participants in MBIs exhibit increases in both mindfulness and self-compassion traits. Multiple metanalyses have also shown that increases in mindfulness and self-compassion are two of the mechanisms by which MBIs lead to decreases in overall stress, anxiety, and depression.

Furthermore, mindfulness meditation could be particularly effective to help POC cope with race-related stress by reducing experiential avoidance. Experiential avoidance is the inability to remain in contact with distressing physical sensations, thoughts, and emotions, even when doing so causes harm in the long term. POC exposed to race-related stressors often develop emotional (e.g., unwillingness to experience sadness after being discriminated against) and behavioral avoidance (e.g., avoiding places where discrimination is likely to occur) that maintain mental health symptoms. As such, mindfulness meditation with its emphasis on bringing awareness to all experiences regardless of their negative valance may serve as an "exposure" strategy that reduces avoidance, leading to decreases in psychological distress.

Considering that rumination (i.e., the passive and repetitive focus on the causes and consequences of one's distress) and emotion suppression (i.e., the active reduction of emotionally expressive behavior when emotionally aroused) are maladaptive emotion regulation strategies often used by POC exposed to race-related stressors, researchers and clinicians have hypothesized that MBIs may be particularly well suited for this population. Research suggests that by cultivating acceptance of and nonjudgmental engagement with thoughts, mindfulness meditation disrupts ruminative tendencies. This hypothesis is consistent with multiple metanalyses showing that the reduction in rumination is a mediator leading to decreases in mental health problems, including stress, anxiety, and depression in MBI programs. In the case of emotion suppression, mindfulness meditation may help individuals identify, describe, and healthy engage with emotions triggered by race-related stressors rather than suppress them, leading to decreases in mental health symptoms. At least one MBI trial has shown that emotion suppression is a significant mediator behind decreases in anxiety and depression among POC. Targeting emotion suppression may be particularly relevant, considering cultural norms and practices among some POC groups (e.g., Asian, Latinx) that encourage down-regulating emotion expression to promote group harmony.

Despite the significant mental health need among individuals who experience discrimination and the existence of promising interventions such as MBIs, POC face numerous barriers to care, including limited access to providers, financial and transportation constraints, as well as stigma. As such, it is not surprising that POC are less likely to seek or receive mental health services compared with their NLW counterparts. Although no single approach will eliminate all barriers driving mental health disparities, the use of technology to provide care could reduce this treatment gap.

Digital interventions have the potential to address the shortage of mental health professionals, mitigate logistic barriers to service utilization, decrease costs associated with EBT implementation, and engage individuals in care who may not seek services otherwise. Among many technological resources available, smartphones represent a promising vehicle for the provision of mental health services. The feasibility of this approach is supported by extensive ownership of mobile devices in the United States. For instance, approximately 81% of Americans have a smartphone, with POC having similar ownership rates as NLW. Compared with NLW, POC are also more likely to be "smartphone dependent" -meaning they rely on these devices to access the internet in the absence of broadband connection at home. Furthermore, POC are also more likely to use their smartphones to seek information about their health than their NLW counterparts. As such, app-based interventions using smartphones may be well-positioned to reach those affected by the digital divide observed in low-income households as these interventions capitalize on already available technology owned by POC.

In addition to their feasibility, there is a growing body of evidence supporting the efficacy of app-based mental health interventions. Although somewhat limited, existing data with POC samples are promising. In the case of app-based MBI, multiple metanalyses show that these interventions are effective in reducing overall stress, anxiety, and depression as well as increasing mindfulness and self-compassion. To the investigators' knowledge, experiential avoidance, rumination, and emotion suppression have not been examined as potential clinical targets in app-based MBIs.

Research Questions and Hypotheses

Aim 1 The purpose of this study is to examine whether this MBI engages relevant mechanisms of change for POC exposed to race-related stress. Based on previous metanalytic studies on mindfulness and self-compassion, the investigators hypothesize that POC who receive the intervention will experience significant increases in both variables compared with POC in the control group. Considering previous studies showing the crucial role of experiential avoidance and emotion suppression, the investigators hypothesize that POC who receive the intervention will experience significant decreases in these three variables compared with POC in the control group.

Aim 2 An additional goal of this study is to test whether POC who receive this MBI experience reductions in mental health symptoms often associated with experiencing race-related stress. Based on previous metanalytic studies, the investigators hypothesize that POC who receive the intervention will experience significant decreases in overall stress, anxiety, and depression compared with POC in the control group.

Aim 3 Related to previous aims, this study will examine whether decreases in the main outcomes of interest (i.e., stress, anxiety, depression) occur via hypothesized mechanisms of change (i.e., mindfulness, self-compassion, experiential avoidance, rumination, emotion suppression). Based on previous metanalytic studies, the investigators hypothesize that the five mechanisms of change examined will be significant mediators leading to decreases in the main outcomes of interest.

Aim 4 This study will also examine app-based MBI acceptability (i.e., extent to which the intervention is agreeable or satisfactory), adherence (i.e., actual use of the intervention), and satisfaction (i.e., positive attitude toward the intervention received) in this high-risk POC population. Considering researchers' and clinicians' concerns regarding potential cultural mismatches between POC's backgrounds and MBIs, the investigators will use both quantitative and qualitative data sources to examine treatment acceptability descriptively. Based on previous studies showing poor treatment engagement in self-directed app-based interventions, the investigators will describe treatment adherence with both behavioral markers and qualitative data. Finally, treatment satisfaction will also be measured using quantitative and qualitative methods. Given that these analyses are descriptive, the investigators do not have specific hypotheses.

ELIGIBILITY:
Inclusion Criteria:

Individuals interested in participating in this study will complete an online screening questionnaire using Qualtrics, a platform that is smartphone compatible. For study inclusion, participants are required to:

1. Identify as a member of a people of color (POC) group
2. Report experiencing elevated levels of race-related stress (i.e., a score of 55 in the IRRS-B or a score of 12 in the MDM)
3. Speak and read English,
4. Not receive psychological services currently
5. Not have practiced mindfulness meditation for more than two hours in the month prior to study commencement
6. Own a smartphone with access to the internet
7. Be willing to install the MBI app and accept daily notifications and text reminders
8. Be at least 18 years old

Screening Measures:

Race-Related Stress. The 22-item Index of Race-Related Stress-Brief (IRRS-B) measures multiple sources of race-related stress, including Individual, Institutional, and Cultural. Participants rate items on a scale ranging from 0 (This Never Happened to Me) to 4 (This Event Happened and I was Extremely Upset), with higher scores indicating more race-related stress. The IRRS-B was developed with a POC sample (i.e., Blacks), showing adequate reliability (α = .78) for both Cultural and Individual subscales and acceptable reliability (α = .69) for the Institutional subscale. For study inclusion, participants need to obtain a score of 55, which represents elevated race-related stress.

Perceived Discrimination. The 8-item Multicultural Discrimination Module (MDM) measures perceived discrimination. Participants rate items on a scale ranging from 1 (Never) to 4 (Often) with higher scores indicating more levels of perceived discrimination. The MDM was developed using a U.S. population-based sample (approximately 40% POC) and has shown good internal consistency (α = .81 - .88) in a previous study. For study inclusion, participants need to obtain a score of 12, which represents the 75th percentile of the population distribution.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Change in stress | Through study completion, 1-2 months
  The 10-item Perceived Stress Scale (PSS) measures stress. Participants rate items on a scale ranging from 0 (Never) to 4 (Very Often) with higher scores indicating more stress. The PSS has shown good reliability (α = .84 - .86) and validity, and it is commonly used in MBI research.
Change in anxiety | Through study completion, 1-2 months
  The General Anxiety Disorder (GAD-7) measures anxiety symptoms. Participants rate items on a scale ranging from 0 (Not at all) to 3 (Nearly Every Day) with higher scores indicating more severe anxiety symptoms. The GAD-7 has shown good internal consistency (α = .89 - .90) and validity in POC samples.
Change in depression | Through study completion, 1-2 months
  The 8-item Patient Health Questionnaire (PHQ-8) measures depressive symptoms. Participants rate items on a scale ranging from 0 (Not at all) to 3 (Nearly Every Day) with higher scores indicating more severe depressive symptoms.The PHQ-8 omits an item assessing suicidal ideation and self-harm included in the original PHQ-9, which makes it more adequate for self-guided digital intervention research. Furthermore, metanalytic work suggests that the PHQ-8 is practically equivalent to the original measure. The PHQ-8 has good reliability (α = .86 - .89) and has shown validity across different racial/ethnic groups.

SECONDARY OUTCOMES:
Change in mindfulness | Through study completion, 1-2 months
  The 15-item Mindful Attention Awareness Scale (MAAS) measures mindfulness trait. Participants rate items using a scale ranging from 1 (Almost Always 1) to 6 (Almost Never) with higher scores indicating more mindfulness. The MAAS has shown good internal consistency (α = .80 - .87) during its development.
Change in self-Compassion | Through study completion, 1-2 months
  The 12-item Self-Compassion Scale, Short Form (SCS-SF) measures self-compassion trait. Participants rate items using a scale ranging from 1 (Almost Never) to 5 (Almost Always) with higher scores indicating more self-compassion. The SCS-SF has shown good internal consistency (α = .86) and validity in a sample with significant POC representation.
Change in experiential avoidance | Through study completion, 1-2 months
  The 15-item Brief Experiential Avoidance Questionnaire (BEAQ) measures experiential avoidance. Participants rate their responses in a scale ranging from 1 (Strongly Disagree) to 6 (Strongly Agree) with higher scores indicating higher experiential avoidance. The BAEQ has shown good internal consistency (α = .80 - .86) and construct validity.
Change in rumination | Through study completion, 1-2 months
  The 5-item Brooding subscale of the short version of the Ruminative Response Scale (RRS-SF) measures rumination. Participants rate their responses in a scale ranging from 1 (Almost Never) to 4 (Almost Always) with higher scores indicating more rumination. The RRS-SF Brooding subscale has shown adequate internal consistency (α = .79) and validity in studies with POC samples that experience discrimination.
Change in emotion suppression | Through study completion, 1-2 months
  The 4-item Expressive Suppression of the Emotion Regulation Questionnaire (ERQ) measures emotion suppression. Participants rate their responses on a scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with higher scores indicating more emotion suppression. The Expressive Suppression subscale of the ERQ has shown an adequate reliability (α = .68 - .76) and validity in samples with significant POC representation.

OTHER OUTCOMES:
Change in acceptability and appropriateness of the intervention | Through study completion, 1-2 months
  The 16-item Attitudes towards Psychological Online Interventions (APOI) measures experiences with digital interventions. Participants rate items on a scale ranging from 1 (Totally Agree) to 5 (Totally Disagree) with higher scores indicating more perceived acceptability and appropriateness. The APOI has shown good reliability (α = .83) and validity in previous studies.
Change in treatment adherence | Through study completion, 1-2 months
  Number of meditations completed, total time meditated in minutes, and number of days with at least one meditation with will be used as behavioral measures of treatment adherence. This information is tracked by the app.
Change in treatment satisfaction | Through study completion, 1-2 months
  The 7-item Satisfaction with Therapy (ST) subscale of the Satisfaction with Therapy and Therapist Scale-Revised (STTS-R) measures treatment satisfaction. Participants rate items on a scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) with higher scores showing more treatment satisfaction. The ST subscale has shown excellent reliability (α = .92) and validity in a digital intervention study with a racially/ethnically diverse sample.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ramos, MA, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acabchuk, R. L., Simon, M. A., Low, S., Brisson, J. M., & Johnson, B. T. (2021). Measuring Meditation Progress with a Consumer-Grade EEG Device: Caution from a Randomized Controlled Trial. Mindfulness, 12(1), 68-81. https://doi.org/10.1007/s12671-020-01497-1
- [Background] Aguilera A, Berridge C. Qualitative feedback from a text messaging intervention for depression: benefits, drawbacks, and cultural differences. JMIR Mhealth Uhealth. 2014 Nov 5;2(4):e46. doi: 10.2196/mhealth.3660. PMID 25373390
- [Background] Aguilera A, Bruehlman-Senecal E, Demasi O, Avila P. Automated Text Messaging as an Adjunct to Cognitive Behavioral Therapy for Depression: A Clinical Trial. J Med Internet Res. 2017 May 8;19(5):e148. doi: 10.2196/jmir.6914. PMID 28483742
- [Background] Aguilera A, Munoz RF. Text Messaging as an Adjunct to CBT in Low-Income Populations: A Usability and Feasibility Pilot Study. Prof Psychol Res Pr. 2011 Dec 1;42(6):472-478. doi: 10.1037/a0025499. PMID 25525292
- [Background] Alkhaldi G, Hamilton FL, Lau R, Webster R, Michie S, Murray E. The Effectiveness of Prompts to Promote Engagement With Digital Interventions: A Systematic Review. J Med Internet Res. 2016 Jan 8;18(1):e6. doi: 10.2196/jmir.4790. PMID 26747176
- [Background] Alsubaie M, Abbott R, Dunn B, Dickens C, Keil TF, Henley W, Kuyken W. Mechanisms of action in mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR) in people with physical and/or psychological conditions: A systematic review. Clin Psychol Rev. 2017 Jul;55:74-91. doi: 10.1016/j.cpr.2017.04.008. Epub 2017 Apr 23. PMID 28501707
- [Background] Baumel A, Muench F, Edan S, Kane JM. Objective User Engagement With Mental Health Apps: Systematic Search and Panel-Based Usage Analysis. J Med Internet Res. 2019 Sep 25;21(9):e14567. doi: 10.2196/14567. PMID 31573916
- [Background] Benish SG, Quintana S, Wampold BE. Culturally adapted psychotherapy and the legitimacy of myth: a direct-comparison meta-analysis. J Couns Psychol. 2011 Jul;58(3):279-89. doi: 10.1037/a0023626. PMID 21604860
- [Background] Beshai S, Bueno C, Yu M, Feeney JR, Pitariu A. Examining the effectiveness of an online program to cultivate mindfulness and self-compassion skills (Mind-OP): Randomized controlled trial on Amazon's Mechanical Turk. Behav Res Ther. 2020 Nov;134:103724. doi: 10.1016/j.brat.2020.103724. Epub 2020 Sep 10. PMID 32942203
- [Background] Biggers A, Spears CA, Sanders K, Ong J, Sharp LK, Gerber BS. Promoting Mindfulness in African American Communities. Mindfulness (N Y). 2020 Oct;11(10):2274-2282. doi: 10.1007/s12671-020-01480-w. Epub 2020 Aug 21. PMID 33584869
- [Background] Bor J, Venkataramani AS, Williams DR, Tsai AC. Police killings and their spillover effects on the mental health of black Americans: a population-based, quasi-experimental study. Lancet. 2018 Jul 28;392(10144):302-310. doi: 10.1016/S0140-6736(18)31130-9. Epub 2018 Jun 21. PMID 29937193
- [Background] Borghouts J, Eikey E, Mark G, De Leon C, Schueller SM, Schneider M, Stadnick N, Zheng K, Mukamel D, Sorkin DH. Barriers to and Facilitators of User Engagement With Digital Mental Health Interventions: Systematic Review. J Med Internet Res. 2021 Mar 24;23(3):e24387. doi: 10.2196/24387. PMID 33759801
- [Background] Brake CA, Sauer-Zavala S, Boswell JF, Gallagher MW, Farchione TJ, Barlow DH. Mindfulness-Based Exposure Strategies as a Transdiagnostic Mechanism of Change: An Exploratory Alternating Treatment Design. Behav Ther. 2016 Mar;47(2):225-38. doi: 10.1016/j.beth.2015.10.008. Epub 2015 Nov 7. PMID 26956654
- [Background] Brondolo E, Brady Ver Halen N, Pencille M, Beatty D, Contrada RJ. Coping with racism: a selective review of the literature and a theoretical and methodological critique. J Behav Med. 2009 Feb;32(1):64-88. doi: 10.1007/s10865-008-9193-0. Epub 2009 Jan 6. PMID 19127420
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Bruehlman-Senecal E, Aguilera A, Schueller SM. Mobile Phone-Based Mood Ratings Prospectively Predict Psychotherapy Attendance. Behav Ther. 2017 Sep;48(5):614-623. doi: 10.1016/j.beth.2017.01.002. Epub 2017 Jan 9. PMID 28711112
- [Background] Bunge E, Cook HM, Bond M, Williamson RE, Cano M, Barrera AZ, Leykin Y, Munoz RF. Comparing Amazon Mechanical Turk with unpaid internet resources in online clinical trials. Internet Interv. 2018 Apr 15;12:68-73. doi: 10.1016/j.invent.2018.04.001. eCollection 2018 Jun. PMID 30135770
- [Background] Carter, E. R., & Murphy, M. C. (2015). Group-based Differences in Perceptions of Racism: What Counts, to Whom, and Why? Social and Personality Psychology Compass, 9(6), 269-280. https://doi.org/10.1111/spc3.12181
- [Background] Carter, R. T., Johnson, V. E., Kirkinis, K., Roberson, K., Muchow, C., & Galgay, C. (2019). A Meta-Analytic Review of Racial Discrimination: Relationships to Health and Culture. Race and Social Problems, 11(1), 15-32. https://doi.org/10.1007/s12552-018-9256-y
- [Background] Castellanos, R., Yildiz Spinel, M., Phan, V., Orengo-Aguayo, R., Humphreys, K. L., & Flory, K. (2020). A Systematic Review and Meta-Analysis of Cultural Adaptations of Mindfulness-Based Interventions for Hispanic Populations. Mindfulness, 11(2), 317-332. https://doi.org/10.1007/s12671-019-01210-x
- [Background] Chae DH, Yip T, Martz CD, Chung K, Richeson JA, Hajat A, Curtis DS, Rogers LO, LaVeist TA. Vicarious Racism and Vigilance During the COVID-19 Pandemic: Mental Health Implications Among Asian and Black Americans. Public Health Rep. 2021 Jul-Aug;136(4):508-517. doi: 10.1177/00333549211018675. Epub 2021 May 25. PMID 34034574
- [Background] Chiesa A, Malinowski P. Mindfulness-based approaches: are they all the same? J Clin Psychol. 2011 Apr;67(4):404-24. doi: 10.1002/jclp.20776. Epub 2011 Jan 19. PMID 21254062
- [Background] Clarke J, Draper S. Intermittent mindfulness practice can be beneficial, and daily practice can be harmful. An in depth, mixed methods study of the "Calm" app's (mostly positive) effects. Internet Interv. 2019 Nov 16;19:100293. doi: 10.1016/j.invent.2019.100293. eCollection 2020 Mar. PMID 31890639
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cook BL, Trinh NH, Li Z, Hou SS, Progovac AM. Trends in Racial-Ethnic Disparities in Access to Mental Health Care, 2004-2012. Psychiatr Serv. 2017 Jan 1;68(1):9-16. doi: 10.1176/appi.ps.201500453. Epub 2016 Aug 1. PMID 27476805
- [Background] Cooper D, Yap K, Batalha L. Mindfulness-based interventions and their effects on emotional clarity: A systematic review and meta-analysis. J Affect Disord. 2018 Aug 1;235:265-276. doi: 10.1016/j.jad.2018.04.018. Epub 2018 Apr 5. PMID 29660642
- [Background] Cotter, E. W., & Jones, N. (2020). A Review of Latino/Latinx Participants in Mindfulness-Based Intervention Research. Mindfulness, 11(3), 529-553. https://doi.org/10.1007/s12671-019-01266-9
- [Background] Craig C, Hiskey S, Spector A. Compassion focused therapy: a systematic review of its effectiveness and acceptability in clinical populations. Expert Rev Neurother. 2020 Apr;20(4):385-400. doi: 10.1080/14737175.2020.1746184. Epub 2020 Apr 10. PMID 32196399
- [Background] Cramer H, Hall H, Leach M, Frawley J, Zhang Y, Leung B, Adams J, Lauche R. Prevalence, patterns, and predictors of meditation use among US adults: A nationally representative survey. Sci Rep. 2016 Nov 10;6:36760. doi: 10.1038/srep36760. PMID 27829670
- [Background] Crandall A, Cheung A, Young A, Hooper AP. Theory-Based Predictors of Mindfulness Meditation Mobile App Usage: A Survey and Cohort Study. JMIR Mhealth Uhealth. 2019 Mar 22;7(3):e10794. doi: 10.2196/10794. PMID 30900992
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Crowe M, Inder M, Porter R. Conducting qualitative research in mental health: Thematic and content analyses. Aust N Z J Psychiatry. 2015 Jul;49(7):616-23. doi: 10.1177/0004867415582053. Epub 2015 Apr 21. PMID 25900973
- [Background] Cummings JR, Allen L, Clennon J, Ji X, Druss BG. Geographic Access to Specialty Mental Health Care Across High- and Low-Income US Communities. JAMA Psychiatry. 2017 May 1;74(5):476-484. doi: 10.1001/jamapsychiatry.2017.0303. PMID 28384733
- [Background] DeLuca, S. M., Kelman, A. R., & Waelde, L. C. (2018). A Systematic Review of Ethnoracial Representation and Cultural Adaptation of Mindfulness- and Meditation-Based Interventions. Psychological Studies, 63(2), 117-129. https://doi.org/10.1007/s12646-018-0452-z
- [Background] Economides M, Martman J, Bell MJ, Sanderson B. Improvements in Stress, Affect, and Irritability Following Brief Use of a Mindfulness-based Smartphone App: A Randomized Controlled Trial. Mindfulness (N Y). 2018;9(5):1584-1593. doi: 10.1007/s12671-018-0905-4. Epub 2018 Mar 1. PMID 30294390
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Fuchs C, Lee JK, Roemer L, Orsillo SM. Using Mindfulness- and Acceptance-Based Treatments With Clients From Nondominant Cultural and/or Marginalized Backgrounds: Clinical Considerations, Meta-Analysis Findings, and Introduction to the Special Series. Cogn Behav Pract. 2013 Feb;20(1):1-12. doi: 10.1016/j.cbpra.2011.12.004. PMID 26294894
- [Background] Fung J, Kim JJ, Jin J, Chen G, Bear L, Lau AS. A Randomized Trial Evaluating School-Based Mindfulness Intervention for Ethnic Minority Youth: Exploring Mediators and Moderators of Intervention Effects. J Abnorm Child Psychol. 2019 Jan;47(1):1-19. doi: 10.1007/s10802-018-0425-7. PMID 29654540
- [Background] Gal E, Stefan S, Cristea IA. The efficacy of mindfulness meditation apps in enhancing users' well-being and mental health related outcomes: a meta-analysis of randomized controlled trials. J Affect Disord. 2021 Jan 15;279:131-142. doi: 10.1016/j.jad.2020.09.134. Epub 2020 Oct 7. PMID 33049431
- [Background] Galante J, Friedrich C, Dawson AF, Modrego-Alarcon M, Gebbing P, Delgado-Suarez I, Gupta R, Dean L, Dalgleish T, White IR, Jones PB. Mindfulness-based programmes for mental health promotion in adults in nonclinical settings: A systematic review and meta-analysis of randomised controlled trials. PLoS Med. 2021 Jan 11;18(1):e1003481. doi: 10.1371/journal.pmed.1003481. eCollection 2021 Jan. PMID 33428616
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474
- [Background] Green CA, Duan N, Gibbons RD, Hoagwood KE, Palinkas LA, Wisdom JP. Approaches to Mixed Methods Dissemination and Implementation Research: Methods, Strengths, Caveats, and Opportunities. Adm Policy Ment Health. 2015 Sep;42(5):508-23. doi: 10.1007/s10488-014-0552-6. PMID 24722814
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Guendelman S, Medeiros S, Rampes H. Mindfulness and Emotion Regulation: Insights from Neurobiological, Psychological, and Clinical Studies. Front Psychol. 2017 Mar 6;8:220. doi: 10.3389/fpsyg.2017.00220. eCollection 2017. PMID 28321194
- [Background] Nagayama Hall GC, Hong JJ, Zane NW, Meyer OL. Culturally-Competent Treatments for Asian Americans: The Relevance of Mindfulness and Acceptance-Based Psychotherapies. Clin Psychol (New York). 2011 Sep 1;18(3):215-231. doi: 10.1111/j.1468-2850.2011.01253.x. PMID 22065893
- [Background] Hall GC, Ibaraki AY, Huang ER, Marti CN, Stice E. A Meta-Analysis of Cultural Adaptations of Psychological Interventions. Behav Ther. 2016 Nov;47(6):993-1014. doi: 10.1016/j.beth.2016.09.005. Epub 2016 Sep 30. PMID 27993346
- [Background] Hanley, A. W., Abell, N., Osborn, D. S., Roehrig, A. D., & Canto, A. I. (2016). Mind the Gaps: Are Conclusions about Mindfulness Entirely Conclusive? Journal of Counseling and Development, 94(1), 103-113. https://doi.org/10.1002/jcad.12066
- [Background] Hawley, L. L., Schwartz, D., Bieling, P. J., Irving, J., Corcoran, K., Farb, N. A. S., Anderson, A. K., & Segal, Z. V. (2014). Mindfulness Practice, Rumination and Clinical Outcome in Mindfulness-Based Treatment. Cognitive Therapy and Research, 38(1), 1-9. https://doi.org/10.1007/s10608-013-9586-4
- [Background] Hayes, A. M., & Feldman, G. (2004). Clarifying the Construct of Mindfulness in the Context of Emotion Regulation and the Process of Change in Therapy. Clinical Psychology: Science and Practice, 11(3), 255-262. https://doi.org/10.1093/clipsy/bph080
- [Background] Hendricks, D. S., Lavery, M. R., Bouillon, L. E., & Gotfried, R. S. (2020). Evaluating the Effectiveness of a Mindfulness App Among Academic Advisors. Journal of Technology in Behavioral Science, 5(2), 149-155. https://doi.org/10.1007/s41347-019-00122-w
- [Background] Hermes ED, Lyon AR, Schueller SM, Glass JE. Measuring the Implementation of Behavioral Intervention Technologies: Recharacterization of Established Outcomes. J Med Internet Res. 2019 Jan 25;21(1):e11752. doi: 10.2196/11752. PMID 30681966
- [Background] Hernandez-Ramos R, Aguilera A, Garcia F, Miramontes-Gomez J, Pathak LE, Figueroa CA, Lyles CR. Conducting Internet-Based Visits for Onboarding Populations With Limited Digital Literacy to an mHealth Intervention: Development of a Patient-Centered Approach. JMIR Form Res. 2021 Apr 29;5(4):e25299. doi: 10.2196/25299. PMID 33872184
- [Background] Hinton, D. E., Pich, V., Hofmann, S. G., & Otto, M. W. (2013). Acceptance and Mindfulness Techniques as Applied to Refugee and Ethnic Minority Populations With PTSD: Examples From "Culturally Adapted CBT." Cognitive and Behavioral Practice, 20(1), 33-46. https://doi.org/10.1016/j.cbpra.2011.09.001
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Huberty J, Eckert R, Larkey L, Kurka J, Rodriguez De Jesus SA, Yoo W, Mesa R. Smartphone-Based Meditation for Myeloproliferative Neoplasm Patients: Feasibility Study to Inform Future Trials. JMIR Form Res. 2019 Apr 29;3(2):e12662. doi: 10.2196/12662. PMID 31033443
- [Background] Huey SJ Jr, Polo AJ. Evidence-based psychosocial treatments for ethnic minority youth. J Clin Child Adolesc Psychol. 2008 Jan;37(1):262-301. doi: 10.1080/15374410701820174. PMID 18444061
- [Background] Jayewardene WP, Lohrmann DK, Erbe RG, Torabi MR. Effects of preventive online mindfulness interventions on stress and mindfulness: A meta-analysis of randomized controlled trials. Prev Med Rep. 2016 Nov 14;5:150-159. doi: 10.1016/j.pmedr.2016.11.013. eCollection 2017 Mar. PMID 28050336
- [Background] Kachan D, Olano H, Tannenbaum SL, Annane DW, Mehta A, Arheart KL, Fleming LE, Yang X, McClure LA, Lee DJ. Prevalence of Mindfulness Practices in the US Workforce: National Health Interview Survey. Prev Chronic Dis. 2017 Jan 5;14:E01. doi: 10.5888/pcd14.160034. PMID 28055821
- [Background] Karekla, M., Kasinopoulos, O., Neto, D. D., Ebert, D. D., Van Daele, T., Nordgreen, T., Höfer, S., Oeverland, S., & Jensen, K. L. (2019). Best Practices and Recommendations for Digital Interventions to Improve Engagement and Adherence in Chronic Illness Sufferers. European Psychologist, 24(1), 49-67. https://doi.org/10.1027/1016-9040/a000349
- [Background] Kazdin, A. E. (2015). Technology-Based Interventions and Reducing the Burdens of Mental Illness: Perspectives and Comments on the Special Series. Cognitive and Behavioral Practice, 22(3), 359-366. https://doi.org/10.1016/j.cbpra.2015.04.004
- [Background] Kazdin AE. Annual Research Review: Expanding mental health services through novel models of intervention delivery. J Child Psychol Psychiatry. 2019 Apr;60(4):455-472. doi: 10.1111/jcpp.12937. Epub 2018 Jun 13. PMID 29900543
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lau, A. (2006). Making the Case for Selective and Directed Cultural Adaptations of Evidence-Based Treatments: Examples From Parent Training. Clinical Psychology: Science and Practice, 13(4), 295-310. https://doi.org/10.1111/j.1468-2850.2006.00042.x
- [Background] Laurie J, Blandford A. Making time for mindfulness. Int J Med Inform. 2016 Dec;96:38-50. doi: 10.1016/j.ijmedinf.2016.02.010. Epub 2016 Mar 2. PMID 26965526
- [Background] Lecomte T, Potvin S, Corbiere M, Guay S, Samson C, Cloutier B, Francoeur A, Pennou A, Khazaal Y. Mobile Apps for Mental Health Issues: Meta-Review of Meta-Analyses. JMIR Mhealth Uhealth. 2020 May 29;8(5):e17458. doi: 10.2196/17458. PMID 32348289
- [Background] Lee RT, Perez AD, Boykin CM, Mendoza-Denton R. On the prevalence of racial discrimination in the United States. PLoS One. 2019 Jan 10;14(1):e0210698. doi: 10.1371/journal.pone.0210698. eCollection 2019. PMID 30629706
- [Background] Leong FT, Kalibatseva Z. Cross-cultural barriers to mental health services in the United States. Cerebrum. 2011 Mar;2011:5. Epub 2011 Mar 23. PMID 23447774
- [Background] Linardon J. Can Acceptance, Mindfulness, and Self-Compassion Be Learned by Smartphone Apps? A Systematic and Meta-Analytic Review of Randomized Controlled Trials. Behav Ther. 2020 Jul;51(4):646-658. doi: 10.1016/j.beth.2019.10.002. Epub 2019 Nov 26. PMID 32586436
- [Background] Linardon J, Cuijpers P, Carlbring P, Messer M, Fuller-Tyszkiewicz M. The efficacy of app-supported smartphone interventions for mental health problems: a meta-analysis of randomized controlled trials. World Psychiatry. 2019 Oct;18(3):325-336. doi: 10.1002/wps.20673. PMID 31496095
- [Background] Linardon J, Fuller-Tyszkiewicz M. Attrition and adherence in smartphone-delivered interventions for mental health problems: A systematic and meta-analytic review. J Consult Clin Psychol. 2020 Jan;88(1):1-13. doi: 10.1037/ccp0000459. Epub 2019 Nov 7. PMID 31697093
- [Background] Littleton H, Grills AE, Kline KD, Schoemann AM, Dodd JC. The From Survivor to Thriver program: RCT of an online therapist-facilitated program for rape-related PTSD. J Anxiety Disord. 2016 Oct;43:41-51. doi: 10.1016/j.janxdis.2016.07.010. Epub 2016 Aug 5. PMID 27513363
- [Background] Martinez JH, Eustis EH, Arbid N, Graham-LoPresti JR, Roemer L. The role of experiential avoidance in the relation between racial discrimination and negative mental health outcomes. J Am Coll Health. 2022 Feb-Mar;70(2):461-468. doi: 10.1080/07448481.2020.1754221. Epub 2020 May 5. PMID 32369427
- [Background] Miller MJ, Keum BT, Thai CJ, Lu Y, Truong NN, Huh GA, Li X, Yeung JG, Ahn LH. Practice recommendations for addressing racism: A content analysis of the counseling psychology literature. J Couns Psychol. 2018 Nov;65(6):669-680. doi: 10.1037/cou0000306. Epub 2018 Aug 9. PMID 30091623
- [Background] Miranda R, Polanco-Roman L, Tsypes A, Valderrama J. Perceived discrimination, ruminative subtypes, and risk for depressive symptoms in emerging adulthood. Cultur Divers Ethnic Minor Psychol. 2013 Oct;19(4):395-403. doi: 10.1037/a0033504. PMID 24188536
- [Background] Mojtabai R, Olfson M, Sampson NA, Jin R, Druss B, Wang PS, Wells KB, Pincus HA, Kessler RC. Barriers to mental health treatment: results from the National Comorbidity Survey Replication. Psychol Med. 2011 Aug;41(8):1751-61. doi: 10.1017/S0033291710002291. Epub 2010 Dec 7. PMID 21134315
- [Background] Neary M, Schueller SM. State of the Field of Mental Health Apps. Cogn Behav Pract. 2018 Nov;25(4):531-537. doi: 10.1016/j.cbpra.2018.01.002. Epub 2018 Mar 5. PMID 33100810
- [Background] Newman, B., Merolla, J. L., Shah, S., Lemi, D. C., Collingwood, L., & Ramakrishnan, S. K. (2020). The Trump Effect: An Experimental Investigation of the Emboldening Effect of Racially Inflammatory Elite Communication. British Journal of Political Science, 1-22. https://doi.org/10.1017/S0007123419000590
- [Background] Oei, T. P. S., & Green, A. L. (2008). The Satisfaction With Therapy and Therapist Scale--Revised (STTS-R) for group psychotherapy: Psychometric properties and confirmatory factor analysis. Professional Psychology: Research and Practice, 39(4), 435-442. https://doi.org/10.1037/0735-7028.39.4.435
- [Background] Olano HA, Kachan D, Tannenbaum SL, Mehta A, Annane D, Lee DJ. Engagement in mindfulness practices by U.S. adults: sociodemographic barriers. J Altern Complement Med. 2015 Feb;21(2):100-2. doi: 10.1089/acm.2014.0269. PMID 25685958
- [Background] Paradies Y, Ben J, Denson N, Elias A, Priest N, Pieterse A, Gupta A, Kelaher M, Gee G. Racism as a Determinant of Health: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 23;10(9):e0138511. doi: 10.1371/journal.pone.0138511. eCollection 2015. PMID 26398658
- [Background] Parkerson HA, Thibodeau MA, Brandt CP, Zvolensky MJ, Asmundson GJ. Cultural-based biases of the GAD-7. J Anxiety Disord. 2015 Apr;31:38-42. doi: 10.1016/j.janxdis.2015.01.005. Epub 2015 Feb 7. PMID 25725310
- [Background] Pascoe EA, Smart Richman L. Perceived discrimination and health: a meta-analytic review. Psychol Bull. 2009 Jul;135(4):531-54. doi: 10.1037/a0016059. PMID 19586161
- [Background] Patel JS, Oh Y, Rand KL, Wu W, Cyders MA, Kroenke K, Stewart JC. Measurement invariance of the patient health questionnaire-9 (PHQ-9) depression screener in U.S. adults across sex, race/ethnicity, and education level: NHANES 2005-2016. Depress Anxiety. 2019 Sep;36(9):813-823. doi: 10.1002/da.22940. Epub 2019 Jul 29. PMID 31356710
- [Background] Proulx J, Croff R, Oken B, Aldwin CM, Fleming C, Bergen-Cico D, Le T, Noorani M. Considerations for Research and Development of Culturally Relevant Mindfulness Interventions in American Minority Communities. Mindfulness (N Y). 2018 Apr;9(2):361-370. doi: 10.1007/s12671-017-0785-z. Epub 2017 Aug 16. PMID 29892321
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Ramos G, Brookman-Frazee L, Kodish T, Rodriguez A, Lau AS. Community providers' experiences with evidence-based practices: The role of therapist race/ethnicity. Cultur Divers Ethnic Minor Psychol. 2021 Jul;27(3):471-482. doi: 10.1037/cdp0000357. Epub 2020 May 11. PMID 32391705
- [Background] Ramos, G., & Chavira, D. A. (2019). Use of Technology to Provide Mental Health Care for Racial and Ethnic Minorities: Evidence, Promise, and Challenges. Cognitive and Behavioral Practice. https://doi.org/10.1016/j.cbpra.2019.10.004
- [Background] Ranganathan P, Pramesh CS, Aggarwal R. Common pitfalls in statistical analysis: Intention-to-treat versus per-protocol analysis. Perspect Clin Res. 2016 Jul-Sep;7(3):144-6. doi: 10.4103/2229-3485.184823. PMID 27453832
- [Background] Rushin, S., & Edwards, G. S. (2018). The Effect of President Trump's Election on Hate Crimes. SSRN Electronic Journal. https://doi.org/10.2139/ssrn.3102652
- [Background] Schmitt MT, Branscombe NR, Postmes T, Garcia A. The consequences of perceived discrimination for psychological well-being: a meta-analytic review. Psychol Bull. 2014 Jul;140(4):921-48. doi: 10.1037/a0035754. Epub 2014 Feb 17. PMID 24547896
- [Background] Schröder, J., Berger, T., Meyer, B., Lutz, W., Hautzinger, M., Späth, C., Eichenberg, C., Klein, J. P., & Moritz, S. (2017). Attitudes Towards Internet Interventions Among Psychotherapists and Individuals with Mild to Moderate Depression Symptoms. Cognitive Therapy and Research, 41(5), 745-756. https://doi.org/10.1007/s10608-017-9850-0
- [Background] Schroder J, Sautier L, Kriston L, Berger T, Meyer B, Spath C, Kother U, Nestoriuc Y, Klein JP, Moritz S. Development of a questionnaire measuring Attitudes towards Psychological Online Interventions-the APOI. J Affect Disord. 2015 Nov 15;187:136-41. doi: 10.1016/j.jad.2015.08.044. Epub 2015 Aug 28. PMID 26331687
- [Background] Schueller, S. M., Hunter, J. F., Figueroa, C., & Aguilera, A. (2019). Use of Digital Mental Health for Marginalized and Underserved Populations. Current Treatment Options in Psychiatry, 6(3), 243-255. https://doi.org/10.1007/s40501-019-00181-z
- [Background] Schumer MC, Lindsay EK, Creswell JD. Brief mindfulness training for negative affectivity: A systematic review and meta-analysis. J Consult Clin Psychol. 2018 Jul;86(7):569-583. doi: 10.1037/ccp0000324. PMID 29939051
- [Background] Shariff-Marco S, Breen N, Landrine H, Reeve BB, Krieger N, Gee GC, Williams DR, Mays VM, Ponce NA, Alegria M, Liu B, Willis G, Johnson TP. MEASURING EVERYDAY RACIAL/ETHNIC DISCRIMINATION IN HEALTH SURVEYS: How Best to Ask the Questions, in One or Two Stages, Across Multiple Racial/Ethnic Groups? Du Bois Rev. 2011 Spring;8(1):159-177. doi: 10.1017/S1742058X11000129. Epub 2011 Apr 15. PMID 29354187
- [Background] Smith JL, Allen JW, Haack C, Wehrmeyer K, Alden K, Lund MB, Mascaro JS. The Impact of App-Delivered Mindfulness Meditation on Functional Connectivity and Self-Reported Mindfulness Among Health Profession Trainees. Mindfulness (N Y). 2021;12(1):92-106. doi: 10.1007/s12671-020-01502-7. Epub 2020 Oct 7. PMID 33052251
- [Background] Smith TB, Rodriguez MD, Bernal G. Culture. J Clin Psychol. 2011 Feb;67(2):166-75. doi: 10.1002/jclp.20757. PMID 21105069
- [Background] Sobczak, L. R., & West, L. M. (2013). Clinical Considerations in Using Mindfulness- and Acceptance-Based Approaches With Diverse Populations: Addressing Challenges in Service Delivery in Diverse Community Settings. Cognitive and Behavioral Practice, 20(1), 13-22. https://doi.org/10.1016/j.cbpra.2011.08.005
- [Background] Sommers-Spijkerman M, Austin J, Bohlmeijer E, Pots W. New Evidence in the Booming Field of Online Mindfulness: An Updated Meta-analysis of Randomized Controlled Trials. JMIR Ment Health. 2021 Jul 19;8(7):e28168. doi: 10.2196/28168. PMID 34279240
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Strohmaier, S., Jones, F. W., & Cane, J. E. (2021). Effects of Length of Mindfulness Practice on Mindfulness, Depression, Anxiety, and Stress: a Randomized Controlled Experiment. Mindfulness, 12(1), 198-214. https://doi.org/10.1007/s12671-020-01512-5
- [Background] Torous J, Nicholas J, Larsen ME, Firth J, Christensen H. Clinical review of user engagement with mental health smartphone apps: evidence, theory and improvements. Evid Based Ment Health. 2018 Aug;21(3):116-119. doi: 10.1136/eb-2018-102891. Epub 2018 Jun 5. PMID 29871870
- [Background] Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Ruminative reconsiderd: A psychometric analysis. Cognitive Therapy and Research, 27(3), 247-259. https://doi.org/10.1023/A:1023910315561
- [Background] Utsey, S. O. (1999). Development and Validation of a Short Form of the Index of Race-Related Stress (IRRS)-Brief Version. Measurement and Evaluation in Counseling and Development, 32(3), 149-167. https://doi.org/10.1080/07481756.1999.12068981
- [Background] van der Velden AM, Kuyken W, Wattar U, Crane C, Pallesen KJ, Dahlgaard J, Fjorback LO, Piet J. A systematic review of mechanisms of change in mindfulness-based cognitive therapy in the treatment of recurrent major depressive disorder. Clin Psychol Rev. 2015 Apr;37:26-39. doi: 10.1016/j.cpr.2015.02.001. Epub 2015 Feb 11. PMID 25748559
- [Background] Vines AI, Ward JB, Cordoba E, Black KZ. Perceived Racial/Ethnic Discrimination and Mental Health: a Review and Future Directions for Social Epidemiology. Curr Epidemiol Rep. 2017 Jun;4(2):156-165. doi: 10.1007/s40471-017-0106-z. Epub 2017 Apr 27. PMID 28920011
- [Background] Waldron, E. M., Hong, S., Moskowitz, J. T., & Burnett-Zeigler, I. (2018). A Systematic Review of the Demographic Characteristics of Participants in US-Based Randomized Controlled Trials of Mindfulness-Based Interventions. Mindfulness, 9(6), 1671-1692. https://doi.org/10.1007/s12671-018-0920-5
- [Background] Williams DR. Stress and the Mental Health of Populations of Color: Advancing Our Understanding of Race-related Stressors. J Health Soc Behav. 2018 Dec;59(4):466-485. doi: 10.1177/0022146518814251. PMID 30484715
- [Background] Zvolensky MJ, Jardin C, Garey L, Robles Z, Sharp C. Acculturative stress and experiential avoidance: relations to depression, suicide, and anxiety symptoms among minority college students. Cogn Behav Ther. 2016 Nov;45(6):501-17. doi: 10.1080/16506073.2016.1205658. Epub 2016 Jul 22. PMID 27448042
- [Background] Wu Y, Levis B, Riehm KE, Saadat N, Levis AW, Azar M, Rice DB, Boruff J, Cuijpers P, Gilbody S, Ioannidis JPA, Kloda LA, McMillan D, Patten SB, Shrier I, Ziegelstein RC, Akena DH, Arroll B, Ayalon L, Baradaran HR, Baron M, Bombardier CH, Butterworth P, Carter G, Chagas MH, Chan JCN, Cholera R, Conwell Y, de Manvan Ginkel JM, Fann JR, Fischer FH, Fung D, Gelaye B, Goodyear-Smith F, Greeno CG, Hall BJ, Harrison PA, Harter M, Hegerl U, Hides L, Hobfoll SE, Hudson M, Hyphantis T, Inagaki M, Jette N, Khamseh ME, Kiely KM, Kwan Y, Lamers F, Liu SI, Lotrakul M, Loureiro SR, Lowe B, McGuire A, Mohd-Sidik S, Munhoz TN, Muramatsu K, Osorio FL, Patel V, Pence BW, Persoons P, Picardi A, Reuter K, Rooney AG, Santos IS, Shaaban J, Sidebottom A, Simning A, Stafford L, Sung S, Tan PLL, Turner A, van Weert HC, White J, Whooley MA, Winkley K, Yamada M, Benedetti A, Thombs BD. Equivalency of the diagnostic accuracy of the PHQ-8 and PHQ-9: a systematic review and individual participant data meta-analysis - ERRATUM. Psychol Med. 2020 Dec;50(16):2816. doi: 10.1017/S0033291719002137. Epub 2019 Aug 19. No abstract available. PMID 31423953
- [Derived] Ramos G, Aguilera A, Montoya A, Lau A, Wen CY, Cruz Torres V, Chavira D. App-Based Mindfulness Meditation for People of Color Who Experience Race-Related Stress: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 14;11(4):e35196. doi: 10.2196/35196. PMID 35436228